CLINICAL TRIAL: NCT06719960
Title: How Are Cognitive Functions Affected by Different Sedation Methods in Geriatric Endoscopic Retrograde Cholangiopancreatography Patients?
Brief Title: How Are Cognitive Functions Affected by Different Sedation Methods in Geriatric Patients?
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-4565
Record Dates: First submitted 2024-11-19; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cognition; Sedation for Gastroenteric Endoscopic Procedure; Geriatric Patients
Keywords: FRAIL; COGNITIVE FUNCTION; ERCP; PROPOFOL; DEXMEDETOMIDINE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol: aged 65 years and older who received propofol
  Interventions: Drug: Propofol group
- Dexmedetomidine: aged 65 years and older who received propofol + dexmedetomidine
  Interventions: Drug: Dexmedetomidine group

INTERVENTIONS:
Drug: Dexmedetomidine group — To evaluate cognitive function, Mini Mental State Examination (MMSE) was administered 3 times before the procedure and 2 hours and 24 hours after the procedure. Frailty level of the patient was determined using the frail frailty questionnaire. Each patient received 0.5µg/kg fentanyl (iv). In the dexmedetomidine group, in addition to propofol infusion at the same doses, dexmedetomidine 0.5 μg/kg-1 loading dose was administered within 10 minutes and then continued as infusion at a dose of 0.2-0.7 μg/kg/h.
  Groups: Dexmedetomidine
Drug: Propofol group — To evaluate cognitive function, Mini Mental State Examination (MMSE) was administered 3 times before the procedure and 2 hours and 24 hours after the procedure. Frailty level of the patient was determined using the frail frailty questionnaire. Each patient received 0.5µg/kg fentanyl (iv). In the propofol group, propofol loading dose: 0.2-0.5mg/kg, maintenance infusion dose: 0.5-4mg/kg/h was continued.
  Groups: Propofol

SUMMARY:
The investigators wanted to observe the change in the level of consciousness of patients undergoing ERCP after anesthesia. For this, the investigators evaluated the patients with the mini mental state examination test and the frail scale.

DETAILED DESCRIPTION:
Background and Aim: For patients, endoscopic retrograde cholangiopancreatography (ERCP) is a painful procedure and requires deeper sedation and less body movement than routine gastrointestinal endoscopy. Different sedation methods can be used during the ERCP procedure, which is increasingly used in elderly patients, but their effects on cognitive functions are not clearly known. The main aim of our study was to observe the effect of different sedation methods routinely used in geriatric ERCP patients on cognitive functions.

Methods: Our observational prospective study included 184 inpatients aged 65 years and older who received propofol or propofol + dexmedetomidine for sedation during ERCP. To evaluate cognitive function, Mini Mental State Examination (MMSE) was administered 3 times before the procedure and 2 hours and 24 hours after the procedure. Frailty level of the patient was determined using the frail frailty questionnaire. Each patient received 0.5µg/kg fentanyl (iv). In the propofol group, propofol loading dose: 0.2-0.5mg/kg, maintenance infusion dose: 0.5-4mg/kg/h was continued. In the dexmedetomidine group, in addition to propofol infusion at the same doses, dexmedetomidine 0.5 μg/kg-1 loading dose was administered within 10 minutes and then continued as infusion at a dose of 0.2-0.7 μg/kg/h. Ramsey score was kept at 3-4. ERCP procedure time, total amount of propofol and dexmedetomidine used, atropine and ephedrine administered additionally were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years older and who underwent ERCP and were hospitalized were included in the study.

Exclusion Criteria:

* Patients with 2nd and 3rd degree Atrioventricular Block,
* Recent history of stroke
* Severe hypotensive
* Cardiorespiratory instability
* Substance abuse
* Psychotic illness
* Severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients processed at Ankara Bilkent City Hospital ERCP unit
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Assesment of cognitive function | Maximum 1 day (Mini Mental State Examination scores can be between 0-30. Less than 10 is considered severe impairment, 10-19 is considered moderate dementia, 19-24 is considered early dementia and 25 and above is considered normal)
  Evaluating patients with Mini Mental State Examination (MMSE). Cognitive disfunctions are recorded

CONTACTS AND LOCATIONS:
Overall Officials: FİLİZ KAYA, MD., Study Chair
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share results after published for one year
Supporting Information: CSR
Time Frame: one year
Access Criteria: Researchers

REFERENCES:
- [Result] Qian XL, Zhang W, Liu MZ, Zhou YB, Zhang JM, Han L, Peng YM, Jiang JH, Wang QD. Dexmedetomidine improves early postoperative cognitive dysfunction in aged mice. Eur J Pharmacol. 2015 Jan 5;746:206-12. doi: 10.1016/j.ejphar.2014.11.017. Epub 2014 Nov 20. PMID 25460022
- [Result] Lei D, Sha Y, Wen S, Xie S, Liu L, Han C. Dexmedetomidine May Reduce IL-6 Level and the Risk of Postoperative Cognitive Dysfunction in Patients After Surgery: A Meta-Analysis. Dose Response. 2020 Feb 5;18(1):1559325820902345. doi: 10.1177/1559325820902345. eCollection 2020 Jan-Mar. PMID 32076394
- [Result] Mei B, Xu G, Han W, Lu X, Liu R, Cheng X, Chen S, Gu E, Liu X, Zhang Y; Perioperative Neurocognitive Disorders (PND) Study Group. The Benefit of Dexmedetomidine on Postoperative Cognitive Function Is Unrelated to the Modulation on Peripheral Inflammation: A Single-center, Prospective, Randomized Study. Clin J Pain. 2020 Feb;36(2):88-95. doi: 10.1097/AJP.0000000000000779. PMID 31714323
- [Result] Sun Z, Shi J, Liu C, Zhang J, Liu Y, Wu Y, Han X, Dai H, Wu J, Bo L, Wang F. The Effect of Low-Dose Dexmedetomidine on Perioperative Neurocognitive Dysfunction in Elderly Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP): A Randomized, Controlled, Double-Blind Trial. Drug Des Devel Ther. 2024 Aug 23;18:3715-3725. doi: 10.2147/DDDT.S470514. eCollection 2024. PMID 39193191

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT06719960/SAP_000.pdf